CLINICAL TRIAL: NCT04272866
Title: Comparing the Bond Strength,Microleakage and the Clinical Performance of Three Different Pit and Fissure Sealants (An in Vitro,in Vivo Study)
Brief Title: Comparing Bond Strength,Microleakage and Clinical Performance of Three Pit and Fissure Sealants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sarah Emad Ali El-Din (Other)
Responsible Party: Sponsor-Investigator, Sarah Emad Ali El-Din, Instructor at pediatric dentistry department faculty of dentistry ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PED 18-9M
Record Dates: First submitted 2020-02-01; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Caries Prevention
Keywords: Caries prevention; Pit and fissure sealant; Clinpro; Triage; Embrace
MeSH Terms: conditions — Van der Woude syndrome | interventions — Clinpro Sealant

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Teeth in this group will be sealed with clinpro sealant
  Interventions: Other: Clinpro sealant
- Group2 (Experimental): Teeth in this group will be sealed with embrace wetbond sealant
  Interventions: Other: Embrace wetbond sealant
- Group3 (Experimental): Teeth in this group will be sealed with triage sealant
  Interventions: Other: Triage sealant

INTERVENTIONS:
Other: Clinpro sealant — Resin based sealant
  Arms: Group 1
Other: Embrace wetbond sealant — Moisture tolerant hydrophilic resin based sealant
  Arms: Group2
Other: Triage sealant — Glass ionomer sealant
  Arms: Group3

SUMMARY:
The aim of the study is :-

1. To evaluate and compare the microleakage of three different fissure sealants(resin-based Clinpro sealant, Moisture tolerant resin-based Embrace WetBond sealant and glass ionomer Fuji Triage sealant) in vitro.
2. To evaluate and compare the bond strength of three different fissure sealants(resin-based Clinpro sealant, Moisture tolerant resin-based Embrace WetBond sealant and glass ionomer Fuji Triage sealant) in vitro.
3. To clinically evaluate and compare the retention of three different fissure sealants(resin-based Clinpro sealant, Moisture tolerant resin-based Embrace WetBond sealant and glass ionomer-based Fuji Triage sealant).
4. To clinically evaluate and compare the caries prevention effect of three different fissure sealants(resin-based Clinpro sealant, Moisture tolerant resin-based Embrace WetBond sealant and glass ionomer-based Fuji Triage sealant).

DETAILED DESCRIPTION:
Total of 60 first permanent molar in male and female children aged between 6-9 years included in this prospective study will be selected randomly from the outpatient Pediatric Dentistry and Dental Public Health Department Faculty of Dentistry Ain Shams University.

Informed consent will be signed for each case by the patient's parent or guardian after thorough explanation of the study.

Procedural Steps:

In vivo

1. Teeth will be divided equally into 3 groups randomly according to the type of sealant used.
2. Pit and fissure sealant application will be conducted by a single operator.
3. A thorough oral prophylaxis of both upper and lower arches was done, followed by polishing using a slurry of pumice and rotating brush to ensure removal of debris from fissures.
4. The occlusal surfaces were then thoroughly cleaned with water to remove all traces of pumice. Isolation of permanent first molars will be obtained using cotton rolls and a saliva ejector.

Group 1(Clinpro sealant)Active control

1. The occlusal surface will be dried and etched with 37% phosphoric acid gel for 30 s
2. Thorough rinsing for 30 s using an oil-free air-water syringe.
3. Clinpro™ Sealant then applied with the brush applicator and light cured for 20 s using visible light cure unit.

Group 2(Embrace WetBond sealant)

1. Etching the teeth for 15 seconds with a phosphoric-acid etchant.
2. Then rinse the etchant from the teeth with an air-water spray for 10 seconds,
3. followed by very light drying of the treated surfaces. With Embrace Wet-Bond, the typical dull, frosted appearance of the etched surface is not desired. Rather, the surface should be lightly dried and very slightly moist with a glossy appearance. To accomplish this, a cotton pellet should be used to remove the excess moisture There should be no visible pooling or drops of water on the tooth surfaces.
4. Applying the Embrace WetBond sealant to the occlusal surface using the supplied applicator tip After dispensing, use a brush applicator to place the sealant, covering all pits and fissures and extending onto the cusp ridges. The final sealant thickness upon application should be at least 0.3 mm.
5. After application, light-cure the sealant for 10 seconds, holding the light-curing probe at right angles to the occlusal surface as close as possible using a high-intensity curing light.

Group 3 (Fuji Triage sealant)

1. The occlusal surfaces conditioned with Dentin Conditioner for 20 s and then rinsed for another 20 s, followed by drying by blotting with a cotton pellet and gently blowing with an air syringe. The surfaces appeared moist and not desiccated.
2. Fuji Triage sealant will then applied to the occlusal surface using a plastic-filling instrument and a disposable nylon brush to spread it into the pits and fissures.
3. The material is self-curing, but a light-curing device can be used for 20 to 40 seconds to hasten setting.
4. When the material loses its glossy appearance, one drop of Fuji Coat is dispensed The coating is applied with a brush to the treated surface and adjacent areas, and light curing is applied .

Articulating paper was used to check the occlusion and any premature contacts were adjusted. The patients were instructed not to eat or drink anything for 30 min, and not to bite or chew on hard substances for the rest of the day. The patients were recalled after a time interval of 1 and 6 months to evaluate the retention and development of caries using Modified Simonsen's criteria.

Criteria for evaluation: (Modified simonsen's criteria) Score 0: No loss of sealant and no evidence of caries Score 1: Partial loss of sealant and no evidence of caries Score 2: Partial loss of sealant and evidence of caries. Score 3: Complete loss of sealant and no evidence of caries Score 4: Complete loss of sealant and evidence of caries. On recall at 3 and 6th month interval, the sealants were evaluated by visual and tactile examination with a sharp probe for retention. The teeth were visually inspected for caries. The data obtained were tabulated and subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1- First permanent molars fully erupted with deep and retentive fissures,free of caries and free of any periapical radiolucency.

  2- Males and Females 3- Age group between 6-9 years 4- Medically free 5- High caries risk children

Exclusion Criteria:

1. Medically compromised children
2. Uncooperative children.
3. Children with abnormalities in occlusion
4. children with abnormal oral habits

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Retention of the sealants | 6 months
  Retention of the sealants will be evaluated according to modified Simon's criteria
Caries prevention effect of the sealants | 6 months
  Caries prevention effects will be evaluated according to modified Simon's criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Alieldin, Principal Investigator — Faculty of dentistry ain shams university
Locations (1):
- Faculty of dentistry ain shams university, Cairo, Egypt